CLINICAL TRIAL: NCT03698734
Title: Effect of Adding Evening Primrose Oil to Misoprostol in Second Trimester Abortion
Brief Title: Evening Primrose Oil Efficacy in Second Trimester Abortion
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Radwa Rasheedy Ali, Principal Investigator, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ASU obstetrics hosp
Record Dates: First submitted 2018-10-04; First posted 2018-10-09 (Actual); Last update posted 2018-10-09 (Actual); Status verified 2018-10

CONDITIONS: Missed Abortion
MeSH Terms: conditions — Abortion, Missed | interventions — evening primrose oil

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Evening primrose oil (Active Comparator)
  Interventions: Drug: Evening primrose oil(EPO)
- placebo (Placebo Comparator)
  Interventions: Drug: Placebo - Cap

INTERVENTIONS:
Drug: Evening primrose oil(EPO) — primiparous women with missed abortion between(13 to 24 weeks) will receive 1 capsule of EPO( 1000mg) in addition to misopristol
  Arms: Evening primrose oil
Drug: Placebo - Cap — primiparous women with missed abortion between(13 to 24 weeks) will receive 1 capsule of placebo in addition to misopristol
  Arms: placebo

SUMMARY:
efficacy of evening primrose oil in shortening the duration of induction in 2nd trimesteric missed abortion

ELIGIBILITY:
Inclusion Criteria:

* Primiparous women

Exclusion Criteria:

* Previous uterine incision( Cs, myomectomy,)
* Contraindications to medical or surgical uterine evacuations (eg, hemodynamically unstable, coagulopathy)
* Evidence of intra-uterine infection
* Rupture of fetal membranes.
* Intrauterine device in place.
* Allergy to prostaglandins or EPO

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-11-01 (Estimated); Primary Completion 2019-11-01 (Estimated); Study Completion 2019-11-01 (Estimated)

PRIMARY OUTCOMES:
duration of medical induction of abortion | up to 1 week
  time needed for complete expulsion of fetus and placenta

CONTACTS AND LOCATIONS:
Locations (1):
- AinShams university maternity hospital, Cairo, Abbassya, Egypt